CLINICAL TRIAL: NCT04680039
Title: Noninvasive Hemodynamic Parameters Measurements as a Tool for Early Warning of Intradialytic Hypotension in Hemodialysis Patients
Brief Title: Early Warning of Intradialytic Hypotension in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PPGESKD001
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hypotension of Hemodialysis
Keywords: Hemodialysis; Intradialytic hypotension; Remote Monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Continuous monitoring — Identifying intradialytic hypotension using a PPG-based wearable monitor

SUMMARY:
In this study, the investigators will monitor patients undergoing hemodialysis treatment with a non-invasive wearable PPG-based device. Measurements will include blood pressure, heart rate, oxygen saturation, stroke volume, cardiac output, cardiac index and systemic vascular resistance, among others. The aim is to diagnose intradialytic hypotension more rapidly than with current noninvasive methods and prevent related poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with EKSD undergoing chronic hemodialysis treatments for > 3 months.
2. Patients must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
3. Patients must satisfy a medical examiner about their fitness to participate in the study.
4. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with an inability to communicate well with the Principal investigator (PI) and staff (i.e., language problem, poor mental development, or impaired cerebral function).
2. Withholding the dialysis session for any reason prior to initiation.
3. Minors under the age of 18.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 adult subjects (≥18 years) with end stage kidney disease (ESKD) undergoing chronic hemodialysis (HD) treatments in Hadassah Ein-Kerem medical center. A patient can participate more than once.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with intradialytic hypotension | Through study completion, an average of 1 year.
  Using a PPG-based non-invasive wearable monitor to allow early detection of intradialytic hypotension

SECONDARY OUTCOMES:
Determining the pathogenesis of intradialytic hypotension | Through study completion, an average of 1 year.
  Continuous monitoring of numerous hemodynamic parameters will allow to determine the pathogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Dean Nachman, MD, Principal Investigator — The Hadassah Ein Kerem Medical Center, Jerusalem, Israel
Locations (1):
- The Hadassah Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided